CLINICAL TRIAL: NCT02934308
Title: Comparison of the Skin Conductance Values and Patient Pain Scores During Minor Procedures in the ICU
Acronym: ICUPAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-66; 2014-A01770-47 (Other: ANSM)
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICU patients (Experimental)
  Interventions: Device: Skin Conductance Monitor

INTERVENTIONS:
Device: Skin Conductance Monitor
  Other Names: monitors skin conductance values

SUMMARY:
Pain in hospitalized patients has received increasing attention, however due to its subjective nature, it has defied objective, quantitative measurements. If a patient is able to communicate, pain may be assessed using standardized sentences, visual analog scales (VAS) or plain numeric scales.When a patient is unable to communicate, a method that would allow the caregiver to continuously monitor patients' pain and alert the provider that the patient may be in pain would be quite useful. The Pain Monitor uses a novel measurement technique of analyzing changes in skin conductance that can be used in patients who are unable to provide a subjective pain score. This study will compare the relationship between the measurements taken by the PainMonitor and pain scores given by communicative patients to evaluate the safety and efficacy of this monitor during planned, routine procedures.

DETAILED DESCRIPTION:
Although pain must be assessed to be treated, it has been challenging to obtain consistent, objective, and quantifiable measurements. The best methods currently available are subjective scales communicated by the patient such as standardized sentences, visual analog scales (VAS), or plain numeric scales. When a patient is unable to communicate, methods used to monitor pain are inadequate. A device that provides an objective assessment of pain in these patients would alert the patient's caregivers that the patient may be in pain and analgesic treatment is indicated.

Various methods (Evans et al, 2013; Kantor, 2014; Isnardon, 2013) have been proposed to monitor patients' reactions to nociceptive stimulation such as:

* changes in heart rate or blood pressure
* changes in microcirculation
* pupillometry
* EEG
* Auditory or somatosensory evoked potentials All of these methods have been found lacking, mostly due to a lack of specificity for pain. Pupillometry is not suitable for long periods of measurement and is sensitive to concomitant treatment (e.g. opioids).

Galvanometry has the potential to provide specific information related to pain in patients who are unable to communicate.

Since sweat glands are the only organs controlled solely by the sympathetic nervous system, there is a reasonable chance that the use of galvanometry can provide a reliable means of assessing pain. There are numerous papers on this topic; searching in PUBmed on the key words "pain" and "skin conductance" results in more than 250 papers (selected references are included in the list below). The PainMonitor system uses galvanometry to monitor changes in skin conductance responses per sec mirroring the number of bursts in the skin sympathetic nerves. This creates a warning for caregivers to assess the potential that the patient is in pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-89 years (inclusive), in an adult ICU
* Patients admitted to the ICU who are able to communicate their pain and anxiety using a VAS
* Patients must be cooperative and not agitated.
* Planned to have a potentially painful procedure

Exclusion Criteria:

* Diagnosed neuropathic disease
* Use of neostigmine within the past 3 hours
* Use of regional anesthesia at the extremity where the device electrodes are placed -

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity with a confidence interval | 1 year
  Sensitivity and specificity with a confidence interval > 80 % when skin conductance responses per sec are > 0.13 and VAS is equal to or greater than 30 mm. This end point will be reached by 100 patients with at least 10 discrete measurements for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, PhD, Principal Investigator — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No